CLINICAL TRIAL: NCT01488838
Title: A Randomized Phase II Study of Adjuvant Concurrent Radiation and Chemotherapy Versus Radiation Alone in Resected High-Risk Malignant Salivary Gland Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Radiation Therapy Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2111-096
Record Dates: First submitted 2011-12-07; First posted 2011-12-08 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2011-12

CONDITIONS: Malignant Salivary Gland Tumors
MeSH Terms: interventions — Cisplatin

ARMS (2):
- Arm 1: (Experimental): Radiation: 60-66 Gy in 2 Gy daily fractions Cisplatin: 40 mg/m2 weekly during radiation for 7 doses
  Interventions: Drug: Cisplatin: 40 mg/m2 weekly during radiation
- Arm 2: (Active Comparator): Radiation: 60-66 Gy in 2 Gy daily fractions
  Interventions: Radiation: Radiation: 60-66 Gy in 2 Gy daily fractions

INTERVENTIONS:
Drug: Cisplatin: 40 mg/m2 weekly during radiation — Cisplatin: 40 mg/m2 weekly during radiation for 7 doses
  Arms: Arm 1:
Radiation: Radiation: 60-66 Gy in 2 Gy daily fractions — Radiation: 60-66 Gy in 2 Gy daily fractions
  Arms: Arm 2:

SUMMARY:
A Randomized Phase II study of Adjuvant Concurrent Radiation and Chemotherapy versus Radiation alone in Resected High-Risk Malignant Salivary Gland Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically proven diagnosis of a malignant major salivary gland tumor of the following histologic subtypes: high grade mucoepidermoid carcinoma, salivary duct carcinoma or high grade adenocarcinoma;
2. Surgical resection with curative intent within 8 weeks prior to registration;
3. Pathologic stage T3-4 or N1-3 or T1-2, N0 with a close (≤1mm) or microscopically positive surgical margin (AJCC, 7th ed.; see Appendix IV); patients must be free of distant metastases based upon the following minimum diagnostic workup:
4. Zubrod Performance Status 0-1; 3.1.5 Age ≥ 18; 3.1.6 CBC/differential obtained within 4 weeks prior to registration, with adequate bone marrow function 3.1.7 Adequate renal and hepatic function within 4 weeks prior to registration 3.1.8 Negative serum pregnancy test within 2 weeks prior to registration for women of childbearing potential; 3.1.9 Women of childbearing potential and male participants who are sexually active must practice adequate contraception during treatment and for 6 weeks following treatment. 3.1.10 Patients must be deemed able to comply with the treatment plan and follow-up schedule.

Exclusion Criteria:

3.2.1 Patients with residual macroscopic disease after surgery; 3.2.2 Patients with salivary gland malignancies originating from the minor salivary glands; 3.2.3 Patients with histologies other than high grade mucoepidermoid carcinoma, high grade adenocarcinoma or salivary duct carcinoma; 3.2.4 Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years (for example, carcinoma in situ of the breast, oral cavity, or cervix are all permissible); 3.2.5 Prior systemic chemotherapy or radiation therapy for salivary gland malignancy; note that prior chemotherapy for a different cancer is allowable; 3.2.6 Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields; 3.2.7 Severe, active co-morbidity, defined as follows: 3.2.7.1 Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months; 3.2.7.2 Transmural myocardial infarction within the last 6 months; 3.2.7.3 Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration; 3.2.7.4 Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration; 3.2.7.5 Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; Note, however, coagulation parameters are not required for entry into this protocol. 3.2.7.6 Acquired Immune Deficiency Syndrome (AIDS) 3.2.7.7 Pre-existing ≥ grade 2 neuropathy; 3.2.7.8 Prior organ transplant. 3.2.8 Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary; 3.2.9 Significant pre-existing hearing loss, as defined by the patient or treating physician.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Acquire preliminary efficacy data comparing postoperative radiotherapy alone to concurrent chemotherapy and radiation using weekly cisplatin. | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- King Faisal Specialist Hospital& Research Center, Riyadh, Saudi Arabia